CLINICAL TRIAL: NCT07280052
Title: Psychological Support Interventions and Their Effect on Quality of Life and Psychological Functioning in Women With Endometriosis: A Randomized Controlled Trial (ENDOPSY)
Brief Title: Psychological Support Interventions for Women With Endometriosis (ENDOPSY)
Acronym: ENDOPSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Université Lyon 2 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL25_0655; 2025-A02054-45 (Other: ID RCB)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Psychological Support; Psychotherapy; Quality of Life; Anxiety; Depression; Emotional Regulation; Women's Health
MeSH Terms: conditions — Endometriosis; Anxiety Disorders; Depression; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Four-arm parallel randomized study evaluating three psychological interventions versus control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CONTROL Group - No Psychological Intervention (No Intervention): Participants receive no structured psychological intervention during the 5-month study period. Usual medical care continues without modification.
- INDIVIDUAL PSYCHOTHERAPY - Individual Psychotherapy (PI) (Other): Individual psychotherapy sessions conducted by trained clinical psychologists. Ten sessions lasting 45 minutes each are delivered every two weeks over a 5-month period. The intervention focuses on emotional experience, psychological support, and associative processes related to endometriosis.
  Interventions: Behavioral: Individual Psychotherapy
- SOCIO-AESTHETIC GROUP THERAPY - Socio-Aesthetic Group Therapy (PG) (Other): Six socio-aesthetic group therapy workshops delivered every two weeks over approximately three months. Sessions last 2 hours each and include skincare, sensory exploration, self-image work, and shared emotional expression. Co-conducted by a socio-esthetician and a psychologist.
  Interventions: Behavioral: Mixed Psychotherapy
- MIXED PSYCHOTHERAPY - Mixed Individual + Group Psychotherapy (PGI) (Other): Combined intervention including two initial individual sessions, alternating individual and group therapy thereafter, and three closing individual sessions. Duration and number of sessions match the individual and group-only interventions.
  Interventions: Behavioral: Socio-Aesthetic Group Therapy

INTERVENTIONS:
Behavioral: Individual Psychotherapy — Ten individual psychotherapy sessions (45 minutes each) delivered every two weeks for 5 months by trained psychologists.
  Arms: INDIVIDUAL PSYCHOTHERAPY - Individual Psychotherapy (PI)
Behavioral: Socio-Aesthetic Group Therapy — Six socio-aesthetic therapy workshops (2 hours each) every two weeks over 3 months, focusing on body image, sensory experience, and emotional expression.
  Arms: MIXED PSYCHOTHERAPY - Mixed Individual + Group Psychotherapy (PGI)
Behavioral: Mixed Psychotherapy — Combined individual and group psychotherapy including alternating sessions and final integrative sessions matching the number and duration of individual and group interventions.
  Arms: SOCIO-AESTHETIC GROUP THERAPY - Socio-Aesthetic Group Therapy (PG)

SUMMARY:
Endometriosis is associated with severe pain, impaired quality of life and significant psychological distress. Psychological support may help improve emotional regulation, mental health, and quality of life in affected women. This randomized controlled trial evaluates the impact of three psychological support interventions-individual psychotherapy, socio-aesthetic group therapy, and a mixed approach combining both-on psychological symptoms and quality of life. Forty participants will be randomized into four parallel arms. The study hypothesis is that psychological support interventions improve psychological functioning and disease-related quality of life compared with no intervention, and that the combined mixed approach may produce greater benefits than the individual or group interventions alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥18 years
* Clinical diagnosis of endometriosis
* Ability to understand and complete psychological evaluations
* Signed written informed consent

Exclusion Criteria:

* Ongoing psychotherapy
* Cognitive, sensory or language impairments preventing participation
* Participation in another interventional clinical study
* Persons under legal protection
* Non-French speakers
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Endometriosis-Related Quality of Life (EHP-30 score) | Baseline (T1) and 5 months (T2)
  Change in the EHP-30 total score between baseline and post-intervention. Higher scores indicate worse quality of life.

SECONDARY OUTCOMES:
Change in Anxiety Symptoms (HADS-A score) | Baseline and 5 months
  Change in anxiety symptoms measured by the Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A) between baseline and T2.
  The HADS-A consists of 7 items scored from 0 to 3, with a total score ranging from 0 to 21.
  Higher scores indicate more severe anxiety symptoms.
Change in Depression Symptoms (HADS-D score) | Baseline and 5 months
  Change in depressive symptoms measured by the Hospital Anxiety and Depression Scale - Depression subscale (HADS-D) between baseline and T2.
  The HADS-D consists of 7 items scored from 0 to 3, with a total score ranging from 0 to 21.
  Higher scores indicate more severe depressive symptoms.
Change in Alexithymia (TAS-20 score) | Baseline and 5 months
  Change in alexithymia measured by the Toronto Alexithymia Scale - 20 items (TAS-20) between baseline and T2.
  The TAS-20 consists of 20 items scored from 1 to 5, with a total score ranging from 20 to 100.
  Higher scores indicate higher levels of alexithymia.
Change in Emotion Regulation (ERQ scores) | Baseline and 5 months
  Change in emotion regulation measured by the Emotion Regulation Questionnaire (ERQ) cognitive reappraisal and expressive suppression subscales between baseline and T2.
  The ERQ includes two subscales:
  Cognitive Reappraisal (6 items; score range 6 to 42)
  Expressive Suppression (4 items; score range 4 to 28)
  Items are scored on a 7-point Likert scale. Higher scores indicate greater use of the corresponding emotion regulation strategy.
Qualitative Themes Emerging From Semi-Structured Interviews | Baseline and 5 months
  Qualitative analysis of thematic content from baseline and final interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud - Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be made publicly available or shared with external researchers.
  This study collects sensitive psychological and health-related data in a small, single-center cohort. Even after de-identification/pseudonymization, the risk of re-identification cannot be sufficiently minimized.
  Study results may be shared in aggregate form (e.g., summary statistics) in publications and presentations.